CLINICAL TRIAL: NCT05698264
Title: A Pilot Study to Understand the Impact of Therapy With Tumour Treating Fields (TTFields) in NSCLC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nir Peled (Other)
Responsible Party: Sponsor-Investigator, Nir Peled, Head of Oncology, Shaare Zedek Medical Center
Organization: Shaare Zedek Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZMC-0216-22
Record Dates: First submitted 2022-11-23; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Non Small Cell Lung Cancer; EGFR Gene Mutation; Immune Checkpoint Inhibitor
Keywords: TTFields; immune checkpoint inhibitor; Non Small Cell Lung Cancer; NSCLC; EGFR Gene Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NSCLC patients with EGFR mutation (Experimental): The cohort A will focus on the clonal evolution in EGFR mutated lung cancer patients by using circulating tumor DNA (ctDNA) analysis of paired baseline and end-of-treatment (EOT) plasma samples. This cohort will be compared to matched EGFR patients previously analyzed by our group.
  Analysis of paired samples from this study will allow a dissection of events acquired through therapy, specifically which component of the combination therapy may be driving selection of the mutations in comparison with the control group without TTFields.
  Interventions: Device: concomitant TTFields treatment device to standard of care EGFR positive NSCLC treatment
- NSCLC patients planned to receive PD-1 inhibitors (Experimental): The cohort B will study the impact of TTField on the profile, activity, and proliferation of peripheral lymphocytes in NSCLC patients receiving PD-1 inhibitors concomitant to TTFields treatment. Lymphocytes will be purified from whole blood samples for the profile, proliferation, and activity analyzed by FACS.
  Interventions: Device: concomitant TTFields treatment device to standard of care anti PD-1 NSCLC treatment

INTERVENTIONS:
Device: concomitant TTFields treatment device to standard of care EGFR positive NSCLC treatment — Concomitant to drug therapy, patients will receive treatment with Tumor Treating Fields (TTFields), generated by the medical device NovoTTF-200T with a recommended duration of minimum 18 h a day. TTFields administered using insulated transducer arrays applied to the skin surrounding the region of a malignant tumor.
  Arms: NSCLC patients with EGFR mutation
Device: concomitant TTFields treatment device to standard of care anti PD-1 NSCLC treatment — Concomitant to drug therapy, patients will receive treatment with Tumor Treating Fields (TTFields), generated by the medical device NovoTTF-200T with a recommended duration of minimum 18 h a day. TTFields administered using insulated transducer arrays applied to the skin surrounding the region of a malignant tumor.
  Arms: NSCLC patients planned to receive PD-1 inhibitors

SUMMARY:
Low intensity, intermediate frequency (100-300 kHz) alternating electric fields, also known as Tumor Treating Fields (TTFields) were found to have a profound inhibitory effect on the growth rate of a variety of human cancer cells. Previous study showed anti-tumor activity in respect of melanoma, glioblastoma (GBM), breast carcinoma and NSCLC cell lines. This study aims to assess the impact of TTFields on NSCLC though the understanding of tumor evolution and peripheral lymphocytes activity and proliferation.

Concomitant to drug therapy, patients will receive treatment with Tumor Treating Fields (TTFields), generated by the medical device NovoTTF-200T with a recommended duration of minimum 18 h a day. TTFields administered using insulated transducer arrays applied to the skin surrounding the region of a malignant tumor.

50 patients will be recruited according to the study design in two cohorts and will receive TTFields therapy: Cohort A: Adult NSCLC EGFR positive mutation. Cohort B: Adult NSCLC patients to be treated with PD-1 inhibitors. The cohort A will focus on the clonal evolution in EGFR mutated lung cancer patients by using circulating tumor DNA (ctDNA) analysis of paired baseline and end-of-treatment (EOT) plasma samples. The cohort B will study the impact of TTField on the profile, activity, and proliferation of peripheral lymphocytes. Lymphocytes will be purified from whole blood samples for the profile, proliferation, and activity analyzed by FACS.

Treatment with TTFields will be administered until progressive disease, unacceptable toxicity1, withdrawal of consent or death. After the end of treatment, the patients will be followed until data cutoff date or 2 years after the last patient had entered the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 years of age and older.
2. Have histologically or cytologically confirmed lung cancer.
3. Documented next generation sequencing assay performed on tumor sample in Clinical Laboratory Improvement Amendments (CLIA)-approved laboratory.
4. Have at least 1 measurable lesion per RECIST v1.1
5. Have life expectancy ≥3 months.
6. Have Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
7. Must provide a signed and dated informed consent indicating that the participants have been informed of all pertinent aspects of the study, including the potential risks, and is willingly participating.
8. Have the willingness and ability to comply with scheduled visits and study procedures.
9. Cohort A, confirmed EGFR mutation.

Exclusion Criteria:

1. Implanted electronic devices (e.g. pacemaker) in the upper torso.
2. Have been diagnosed with another primary malignancy within the past 3 years (except for adequately treated non-melanoma skin cancer, cervical cancer in situ or prostate cancer, which are allowed within 3 years).
3. Have any condition or illness that, in the opinion of the investigator, would compromise participants' safety or interfere with the evaluation.
4. Be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-20 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Molecular ctDNA characterization under concomitant TTFields therapy - cohort A (EGFR) | 5 years
  The primary outcome measure will be the rate of new somatic mutation detection in circulating tumor DNA (ctDNA) using Next Generation Sequencing (NGS) in patients receiving concurrent TTFields therapy. The measure will be reported as the percentage of patients showing new somatic mutations upon progression of their disease following TTFields treatment.
In vitro peripheral lymphocytes activity characterization under concomitant TTFields therapy - cohort B (under PD-1 inhibitors treatment) | 5 years
  The primary outcome measure will be the evaluation of the impact of combining PD-1 inhibitors with TTFields therapy on peripheral lymphocyte activity using an in vitro assay. Whole blood samples will be collected and the assay will involve the isolation, activation, and labeling of peripheral lymphocytes from patients in cohort B with a panel of antibodies. The analysis will be performed using flow cytometry (FACS) and the longitudinal changes in peripheral lymphocyte activity will be correlated with each patient's response.
Characterization of the impact of TTFields on peripheral lymphocytes proliferation ex-vivo - cohort B (PD-1 inhibitors treatment) | 5 years
  The primary outcome measure will be the quantification of peripheral lymphocyte proliferation in patients receiving PD-1 inhibitors therapy using an in vitro assay. Whole blood samples will be collected and the assay will involve the isolation, labeling, and analysis of peripheral lymphocytes with carboxyfluorescein diacetate succinimidyl ester (CFSE). Proliferation will be measured using flow cytometry (FACS) and the longitudinal changes in peripheral lymphocyte proliferation will be correlated with each patient's response to the therapy in cohort B.

SECONDARY OUTCOMES:
Safety will be assessed by recording adverse events in both cohorts. | 5 years
  Grading of an Adverse Event. The descriptions and grading scales found in the revised NCI Common Toxicity Criteria (CTC) version 4.0 will be utilized for assessing severity of adverse events. If the toxicity is not characterized adequately by the NCI toxicity scale, the investigator will use the adjectives MILD, MODERATE, SEVERE to describe the maximum intensity of the adverse event.
Objective response rate | 5 years
  Objective response rate (ORR) assessed by the investigator, defined as the proportion of the participants with confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid tumors (RECIST) v1.1, after initiation of study treatment.
DoR | 5 years
  Duration of response, defined as the time interval from the time that the measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that the progressive disease is objectively documented or death. Patients without progressive disease or death will be censored at the last valid response assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No